CLINICAL TRIAL: NCT00433095
Title: Vinorelbine (Oral) Plus Trastuzumab for 1st-line Treatment of HER2/Neu Overexpressing Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mamma-2-2004
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2007-02

CONDITIONS: Carcinoma Breast Stage IV
Keywords: Navelbine; Herceptin; oral; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Trastuzumab

INTERVENTIONS:
Drug: Navelbine
Drug: Herceptin
Drug: Navelbine (oraly)

SUMMARY:
1st-line treatment of HER2/neu overexpressing breast cancer

DETAILED DESCRIPTION:
The combination of vinorelbine and trastuzumab was demonstrated to be highly effective in several trials showing response rates in the range of 59-78%. This combination is characterized by good tolerability and can be applied for a prolonged period without the risk of major cumulative toxicity The availability of oral vinorelbine promises a further simplification of therapy. The present trial therefore investigates the safety and efficacy of a combined treatment with trastuzumab and oral vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, metastatic breats cancer.
* HER2-neu overexpression (IHC3+ or IHC2+/FISH+)
* Written informed consent
* no previous therapy with vinorelbine or trastuzumab
* Age * 18 and * 75 years
* Karnofsky-Performance status > 70%
* Life expectance 16 weeks and more
* Availability of at least one target lesion according to RECIST-criteria. Target lesions need to be outside of radiation fields. Bone metastases are excluded as indicator leasions
* Exclusion of pregnancy and adequte contraception during childbearing age.

  * Adequate hematological, renal, and hepatic function
* Normal cardiac function. LVEF should not be >10% below normal.
* Adequate compliance to perform treatment and subsequent follow-up visits

Exclusion Criteria:

* Locoregional recurrence of breast cancer only or development of contralateral breast cancer
* Pregnancy or lactation
* Symptomatic brain- or meningeal metastasis
* Concurrent endocrine antitumor therapy
* Other malignancies except basal cell cancer of the skin or in-situ carcinoma of the cervix
* Peripheral neuropathy >= NCI CTC Grade 2.
* other severel disease which preclude adequate treatment
* Participation in a clinical trial within the last 30 days.
* Psychological, familial, sociological or geographical conditions which preclude treatment according to the protocol or the planned follow-up

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Time to tumor progression
Overall survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, PhD, MD, Principal Investigator — University of Munich - Klinikum Grosshadern; Hans-Joachim Stemmler, PhD, MD, Study Chair — University of Munich - Klinikum Grosshadern
Locations (1):
- University of Munich - Klinikum Grosshdern, Munich, Germany